CLINICAL TRIAL: NCT05923996
Title: Fractional Carbon Dioxide Laser Versus Microbotox Injection in the Treatment of Wide Facial Pores: A Split Face Comparative Study
Brief Title: Fractional Co2 Laser Versus Microbotox Injection in the Treatment of Wide Facial Pores: A Split Face Comparative Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Alaa Eldin Ibrahim, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: treatment of wide facial pores
Record Dates: First submitted 2023-03-14; First posted 2023-06-29 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Skin Abnormalities
MeSH Terms: conditions — Skin Abnormalities | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbotox injection (Experimental): 21 Egyptian patients with wide facial pores will be treated in a split-face manner. In this side of the face will received single session of microbotox injection contains 20 units of botulinum toxin A.
  Interventions: Drug: microbotox
- Fractional carbon dioxide laser in second side of the face (Experimental): 21 Egyptian patients with wide facial pores will be treated in a split-face manner. In this side will be treated by Two sessions of the fractional CO2 laser on this side of the face at 4-weeks intervals.
  Interventions: Radiation: fractional carbon dioxide laser

INTERVENTIONS:
Drug: microbotox — Will be treated by single session of microbotox injection
  Other Names: botulinum toxin type A
  Arms: Microbotox injection
Radiation: fractional carbon dioxide laser — Two sessions of the fractional CO2 laser on this side of the face at 4-weeks intervals
  Arms: Fractional carbon dioxide laser in second side of the face

SUMMARY:
1. Evaluation of fractional Co2 laser as a treatment option for wide pores in skin type (III - VI)
2. Evaluation of mesobotox as a new modality for improving wide pores appearance.
3. Comparison of both treatment modalities in treatment of enlarged pores.

DETAILED DESCRIPTION:
Skin pores (SP), as they are called by laymen, are common and benign features mostly located on the face (nose, cheeks, etc) that generate many aesthetic concerns or complaints.

Enlarged skin pores refer to conditions that present with visible topographic changes of skin surfaces. Although not a medical concern, enlarged pores are a cosmetic concern for a large number of individuals.

Enlarged facial pores affect individuals of different ages, sexes, and races for which many seek treatment. The exact patho-mechanism of enlarged facial pores is not completely understood. Possible causes include genetic predisposition, seborrhea, aging, increased ultraviolet exposure and comedogenic products.

The treatment of dilated facial pores is difficult, and the ideal modality is not established yet. Many treatment modalities reduce facial pores' count and area, including oral and topical medications as well as different wavelengths of laser. Different ablative and non ablative lasers have been used in the treatment of dilated pores with variable outcomes.

The short-term results showed that treatment with low energy level CO2 fractional laser therapy could be a safe and effective option for patients with Fitzpatrick skin Types III and IV who are concerned with enlarged pores.

Microbotox also called mesobotox, is the injection of multiple microdroplets of diluted onabotulinum toxin A into the upper dermis. It has been previously used in study to decrease pore size and to improve skin texture.

Microbotox has been proved to be effective in improving the sheen and texture of the skin, as well as decreasing sweat and sebum production and enlarged pores as it causes atrophy of sebaceous glands, which subsequently causes tightening of the skin envelope.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with wide facial pores any grade.
2. Sex: male and female patient.
3. Age groups: patient above 18 and below 45 years old.
4. Co-operative patient.

Exclusion Criteria:

1. Patient below 18 and above 45 years old.
2. Patient with systemic illness or other dermatological disease.
3. Patient who receive topical treatment for facial wide pores in past month.
4. Patient who receive systemic treatment for facial wide pores in past 2 month.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
pore score | three months
  evaluation of facial pores after four weeks of second session by pore score: score "0" referred to absence of visible pores. score "1" referred to patients with visible pores. score "2" referred to patient with enlarged pores. score "3" referred to patient with black heads when embedded on facial pores.
sebum score | three months
  evaluation the degree of seborea after four weeks of second session by sebum score: 0 (dry skin)
  1. (mild oiliness)
  2. (moderate oiliness)
  3. (severe oiliness)
Quartile improvement scale | three months
  assessment the improvement after four weeks of first session and after four weeks of second session by Quartile improvement scale: 0 = No improvement
  1. = Minor/mild improvement (1%-25%)
  2. = Moderate improvement (26%-50%)
  3. = Marked improvement (51%-75%)
  4. = Very significant improvement (76%-100%)

SECONDARY OUTCOMES:
Likert satisfaction scale | three months
  1. = Very dissatisfied
  2. = Dissatisfied
  3. = Neither satisfied
  4. = Satisfied
  5. = Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Dalia A Ahmed, professor, Study Director — Assiut University; Howida O Mahmoud, lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flament F, Francois G, Qiu H, Ye C, Hanaya T, Batisse D, Cointereau-Chardon S, Seixas MD, Dal Belo SE, Bazin R. Facial skin pores: a multiethnic study. Clin Cosmet Investig Dermatol. 2015 Feb 16;8:85-93. doi: 10.2147/CCID.S74401. eCollection 2015. PMID 25733918
- [Background] Lee SJ, Seok J, Jeong SY, Park KY, Li K, Seo SJ. Facial Pores: Definition, Causes, and Treatment Options. Dermatol Surg. 2016 Mar;42(3):277-85. doi: 10.1097/DSS.0000000000000657. PMID 26918966
- [Background] Tarek E, Mostafa WZ, Allam RSHM, El-Samanoudy SI, Saadi DG. Short-pulsed and Q-switched ND-YAG laser with topical carbon versus fractional CO2 laser in the treatment of enlarged facial pores: A split-face comparative study. Lasers Surg Med. 2022 Feb;54(2):237-244. doi: 10.1002/lsm.23454. Epub 2021 Jul 13. PMID 34255869
- [Background] Eldeeb F, Wahid RM, Alakad R. Fractional carbon dioxide laser versus carbon-assisted Q-switched Nd: YAG laser in the treatment of dilated facial pores. J Cosmet Dermatol. 2021 Dec;20(12):3917-3923. doi: 10.1111/jocd.14311. Epub 2021 Jul 1. PMID 34169628
- [Background] Kwon HH, Choi SC, Lee WY, Jung JY, Park GH. Clinical and Histological Evaluations of Enlarged Facial Skin Pores After Low Energy Level Treatments With Fractional Carbon Dioxide Laser in Korean Patients. Dermatol Surg. 2018 Mar;44(3):405-412. doi: 10.1097/DSS.0000000000001313. PMID 28902036
- [Background] Ahmed El Attar Y, Nofal A. Microbotox for the treatment of wide facial pores: A promising therapeutic approach. J Cosmet Dermatol. 2021 May;20(5):1361-1366. doi: 10.1111/jocd.13675. Epub 2020 Sep 27. PMID 32799408
- [Background] Salem RM, Salah SAE, Ibrahim SE. Microbotox injection versus its topical application following microneedling in the treatment of wide facial pores: A split face comparative study. J Cosmet Dermatol. 2023 Apr;22(4):1249-1255. doi: 10.1111/jocd.15590. Epub 2023 Jan 6. PMID 36606384
- [Background] Sayed KS, Hegazy R, Gawdat HI, Abdel Hay RM, Ahmed MM, Mohammed FN, Allam R, Fahim A. The efficacy of intradermal injections of botulinum toxin in the management of enlarged facial pores and seborrhea: a split face-controlled study. J Dermatolog Treat. 2021 Nov;32(7):771-777. doi: 10.1080/09546634.2019.1708241. Epub 2020 Jan 3. PMID 31865815
- [Background] Saedi N, Petrell K, Arndt K, Dover J. Evaluating facial pores and skin texture after low-energy nonablative fractional 1440-nm laser treatments. J Am Acad Dermatol. 2013 Jan;68(1):113-8. doi: 10.1016/j.jaad.2012.08.041. Epub 2012 Oct 23. PMID 23098639